CLINICAL TRIAL: NCT01809002
Title: A Multicenter, Prospective, Randomized, Subject and Evaluator Blinded Comparative Study of Nerve Cuffs and Avance® Nerve Graft Evaluating Recovery Outcomes for the Repair of Nerve Discontinuities
Brief Title: Comparison of Processed Nerve Allograft and Collagen Nerve Cuffs for Peripheral Nerve Repair
Acronym: RECON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANG-CP-007
Record Dates: First submitted 2013-03-04; First posted 2013-03-12 (Estimated); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Nerve Discontinuities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Processed Nerve Allograft (Experimental): Processed Nerve Allograft
  Interventions: Biological: Processed Nerve Allograft (human)
- Collagen Nerve Cuff (Active Comparator)
  Interventions: Device: Collagen Nerve Cuff

INTERVENTIONS:
Biological: Processed Nerve Allograft (human)
  Arms: Processed Nerve Allograft
Device: Collagen Nerve Cuff — Bovine collagen based nerve cuff
  Arms: Collagen Nerve Cuff

SUMMARY:
Processed Nerve Allograft and Collagen Nerve Cuffs will be compared to assess safety and functional outcomes for the repair of nerve injuries in the hand.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Nerve Injury

Exclusion Criteria:

* Peripheral Neuropathy
* Allergic to Bovine products such as Bovine Collagen Nerve Cuff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Isaacs, MD, Principal Investigator — Virginia Commonwealth University Medical Center; L. Scott Levin, MD FACS, Principal Investigator — University of Pennsylvania
Locations (21):
- United States (21):
  - University California, Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Florida Orthopaedic Institute, Tampa, Florida
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Curtis National Hand Center, Baltimore, Maryland
  - Spectrum Health, Grand Rapids, Michigan
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Hand Surgery Specialists of Nevada, Las Vegas, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Penn State Universtiy, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rothman Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Univeristy of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Marshall Orthopaedics, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isaacs J, Eswaran S, Ilyas A, Means KR, Levin LS. Digital Nerve Repair With Flexor Tendon Injury: Conduits are Less Effective. Hand (N Y). 2025 Dec 30:15589447251406917. doi: 10.1177/15589447251406917. Online ahead of print. PMID 41472406

RESULTS

PARTICIPANT FLOW:
Groups:
- Processed Nerve Allograft: Processed Nerve Allograft
  Processed Nerve Allograft (human)
Period: Overall Study
Arm/Group | Processed Nerve Allograft | Collagen Nerve Cuff
Started | 112 | 108
Completed | 91 | 92
Not Completed | 21 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Processed Nerve Allograft | Collagen Nerve Cuff | Total
Number analyzed (Participants) | 112 | 108 | 220
Age, Continuous [Median (Standard Deviation); unit: Years] — All subjects were randomized.
  Years | 37.2 (13.6) | 39.8 (14.1) | 38.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects were randomized.
  Participants
    Female | 34 | 31 | 65
    Male | 78 | 77 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All subjects were randomized.
  Participants
    Hispanic or Latino | 10 | 16 | 26
    Not Hispanic or Latino | 102 | 90 | 192
    Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — All subjects were randomized.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 17 | 16 | 33
    White | 89 | 85 | 174
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants] — All subjects were randomized.
  participants
    United States | 112 | 108 | 220

OUTCOME MEASURES:

1. Primary Outcome: Static Two-Point Discrimination (Pre-defined Mixed Modeling Approach)
Description: Static two-point discrimination (s2PD) is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm (best case scenario value possible) and 15mm. The failure to respond to stimulus was pre-defined as the worst case scenario value possible (16mm). Missing or incomplete assessments were imputed as the worst case scenario value possible (16mm). Missing or incomplete data was extrapolated using a pre-defined repeated measures mixed modeling approach for calculations in this analysis. This analysis was completed on the Per Protocol population, defined as subjects with at least 6 months follow-up and no major protocol violations.
Time Frame: Month 12
Population: This is the Per Protocol population which includes all patients in baseline population who have completed a minimum of 6 months follow-up and have no major protocol violations. The analysis was performed using a pre-defined statistical analysis with a non-response/failure assigned a worst-case scenario value of 16mm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimeters
Groups:
- Processed Nerve Allograft (PNA): Commercially available Processed Nerve Allograft for repair of nerve gap
- Collagen Nerve Cuff: Commercially available collagen nerve cuff for repair of nerve gap
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 91 | 92
Millimeters | 9.1 [8.116 to 10.041] | 9.3 [8.403 to 10.240]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; The analysis was performed using a pre-defined standard statistical analysis with a non-response/failure assigned a worst-case scenario value of 16mm; Test type: Non-Inferiority — The primary endpoint tested non-inferiority as compared to collagen nerve cuff and superior to no treatment. Non-inferiority is defined as the lower limit of the 95% CI about the difference of > -2 and the upper limit of the 95% CI for s2PD for Avance of < 13 in ITT table; ANCOVA; Mean Difference (Net) = .2, 95% CI 2-sided [-1.087 to 1.574]

2. Primary Outcome: Static Two-Point Discrimination (Data As-reported)
Description: s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm (best case scenario value possible) and 15mm. The failure to respond to stimulus was pre-defined as the worst case scenario value possible (16mm). Missing or incomplete assessments were not imputed. This analysis was completed on the Per Protocol population, defined as subjects with at least 6 months follow-up and no major protocol violations. Data used for this analysis was from 6 months post-surgical follow-up to the date of each subject's latest completed s2PD assessment, whichever came last, assessed up to 12 months.
Time Frame: Up to Month 12
Population: No interpolated data or modeling was used for this analysis. Results by length of nerve gap (gap 5-14mm vs. gap 15-25mm). As there is no pre-defined numerical value for absent response/failure in as-reported data, 'absent' results were not included in this analysis. This is the Per Protocol population which includes all patients in baseline population who have completed a minimum of 6 months follow-up and have no major protocol violations.
Measure: Mean (Full Range); unit: Millimeters
Groups:
- Processed Nerve Allograft (PNA) (Gap 5-14mm); Processed Nerve Allograft (PNA) (Gap 15-25mm): Commercially available Processed Nerve Allograft for repair of nerve gap
- Collagen Nerve Cuff (Gap 5-14mm); Collagen Nerve Cuff (Gap 15-25mm): Commercially available collagen nerve cuff for repair of nerve gap
Arm/Group | Processed Nerve Allograft (PNA) (Gap 5-14mm) | Collagen Nerve Cuff (Gap 5-14mm) | Processed Nerve Allograft (PNA) (Gap 15-25mm) | Collagen Nerve Cuff (Gap 15-25mm)
Number analyzed (Participants) | 56 | 59 | 35 | 33
Millimeters | 7.3 [3 to 14] | 7.5 [2 to 15] | 6.1 [2 to 14] | 7.5 [5 to 14]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) (Gap 15-25mm) vs Collagen Nerve Cuff (Gap 15-25mm); Test type: Superiority; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Processed Nerve Allograft (PNA) (Gap 5-14mm) vs Collagen Nerve Cuff (Gap 5-14mm); Test type: Superiority; p = 0.365, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Response Rate for Recovery of s2PD at Month 12 (Data As-Reported)
Description: This is the percentage of subjects who achieved sensibility as defined by s2PD 2mm-15mm at Month 12. s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. The failure to respond to stimulus was pre-defined as the worst case scenario value possible (16mm). Missing or incomplete assessments were imputed as the worst case scenario value possible (16mm). This analysis was completed on the Intent-to-Treat population, defined as all subjects who were randomized.
Time Frame: Month 12
Population: This is the Intent To Treat population which includes all subjects that were randomized and have a reported value at Month 12. The analysis was performed using a pre-defined statistical analysis with a non-response/failure assigned a worst-case scenario value of 16mm. Missing or incomplete data was not included in this analysis of response rate.
Measure: Number; unit: % of subjects with recovery of s2PD
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 71 | 79
% of subjects with recovery of s2PD | 77.5 | 77.2
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Responders were defined as subjects achieving s2PD of 2-15 mm on the target nerve repair; Test type: Superiority; p = 0.915, Regression, Logistic — The number and percentage of all treated subjects who recovered s2PD in the target repair at Month 12 (i.e., s2PD of 2 - 15 mm) were summarized by repair type. Differences between the repair types were assessed using a logistic regression analysis

4. Secondary Outcome: Percent Recovery to Pre-Injury Baseline (Contralateral Control Value) s2PD at Month 12 (Pre-defined Modeling Approach)
Description: This is the ratio of sensibility at Month 12 relative to sensibility at baseline for which the contralateral control value at Month 12 was used, expressed as a percentage. Pre-injury baseline was defined as s2PD at Month 12 in the contralateral digit associated with the target digit. Percent recovery to Pre-Injury Baseline was defined as: change from Pre-Injury Baseline (Contralateral control value) divided by the Pre-Injury Baseline Value *100. s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. The failure to respond to stimulus was pre-defined as the worst case scenario value possible (16mm). Missing or incomplete assessments were imputed as the worst case scenario value possible (16mm). This analysis was completed on the Intent-to-Treat population, defined as all subjects who were randomized.
Time Frame: Month 12
Population: This is the Intent To Treat population which includes all subjects that were randomized and have a reported value at Month 12. The analysis was performed using a pre-defined statistical analysis with a non-response/failure assigned a worst-case scenario value of 16mm. Missing or incomplete data was extrapolated using a pre-defined repeated mixed measures modeling approach for calculations in this analysis.
Measure: Mean (Full Range); unit: % recovery
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 71 | 79
% recovery | 54.46 [12.5 to 200.0] | 51.67 [18.8 to 150.0]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; ANCOVA — Pre-injury baseline was defined as s2PD in the contralateral digit associated with the target digit; This analysis was assessed in the ITT population, at Month 12 using the LS Mean differences from a repeated measures ANCOVA model; LS Means difference = -2.84, 95% CI 2-sided [-11.6316 to 5.9541]

5. Secondary Outcome: Time to Recovery of s2PD (Data As-reported)
Description: Time to recovery of s2PD was defined as the number of months from Operative day to the return of sensory function (defined as Medical Research Council sensory function score of S3+ or greater) at Month 3, Month 6, Month 9, or Month 12. s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. S4 is s2PD of 2-6mm and S3+ is s2PD of 7-15mm. Those without S3+ and absent values were considered not recovered. This is the Intent To Treat population which includes all subjects that were randomized. Any subject with a value of s2PD of absent was considered not recovered and was therefore not included in this analysis.
Time Frame: Assessed at Month 3, Month 6, Month 9, Month 12 (some patients were seen for their 12-month visit up to 15 calendar months post-op)
Population: This is the Intent To Treat population which includes all subjects that were randomized. Any subject with a value of s2PD of absent was considered not recovered and was therefore not included in this analysis.
Measure: Mean (Full Range); unit: Months
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 112 | 108
Months | 8.0 [3 to 15] | 7.8 [3 to 15]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; p = 0.792, Kaplan-Meier median and 95% CI; Differences between the repair types were assessed with a KM log-rank test that was appropriate for the handing of interval-censored data

6. Secondary Outcome: Medical Research Council (MRC) Classification for Sensory Function Scores at Month 12 (Data As-reported)
Description: MRC classification score is a functional recovery classification. For nerves with sensory targets, outcomes resulting from static two-point discrimination and Semmes-Weinstein Monofilament pressure threshold testing are used to determine the classification score. Sensibility testing for the target repair was performed by a blinded assessor using a standardized discriminator tool and Semmes-Weinstein monofilaments. Upper bound response for static two-point discrimination was 15mm. This is the Intent To Treat population which includes all subjects that were randomized and have a reported value at Month 12. Scale range: Minimum S0 = 0 (no sensibility), S1=1, S2=2, S3=3, S3+=4, maximum S4 = 5 (normative levels of sensibility). Higher values represented better outcomes.
Time Frame: Month 12
Population: This is the Intent To Treat population which includes all subjects that were randomized and have a reported value at Month 12. In this analysis of Month 12 data, MRCC scores are assigned numeric values: S0=0, S1=1, S2=2, S3=3, S3+=4, S4=5.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 71 | 79
Score on a scale | 4.0 [0 to 5] | 4.0 [0 to 5]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; p = 0.526, Wilcoxon (Mann-Whitney); This analysis was completed to detect a distribution shift of the MRCC score between repairs with PNA and repairs with nerve cuff at Month 12

7. Secondary Outcome: Change in Pain Visual Analogue Scale (VAS) Scores at Month 12 (Pre-defined Modeling Approach)
Description: The Visual Analog Scale (VAS) For Pain is a patient reported outcomes scale whereby the patient indicated their current pain level by making a mark on a continuous horizontal 10 centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the subject is currently experiencing. VAS for Pain data were recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing no pain and 100 millimeters representing "the worst pain imaginable". This is the Intent To Treat population which includes all subjects that were randomized. The analysis was performed using a standard statistical analysis on Month 12 data. Missing or incomplete data was extrapolated using a pre-defined repeated measures modeling approach for calculations in this analysis.
Time Frame: Month 12
Population: This is the Intent To Treat population which includes all subjects that were randomized. The analysis was performed using a standard statistical analysis on Month 12 data. The analysis compared Month 12 VAS to Baseline VAS within-group. No between-group analyses were conducted.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 74 | 80
Units on a scale | -24.09 [-100.0 to 50.0] | -24.94 [-100.0 to 50.0]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA); This analysis compares the change in 12 Month Pain VAS scores from Baseline. Missing or incomplete data was extrapolated using a pre-defined repeated measures modeling approach for calculations in this analysis. This analysis assesses each treatment group for clinically meaningful improvement in VAS from Baseline assuming a Meaningful Clinically Important Difference delta of 20 points (mm); Test type: Other; Mean Difference (Final Values) = -24.09

8. Other Pre Specified Outcome: Number of Participants With Persistent and Unresolved Pain (Data As-reported)
Description: No interpolated data or modeling was used for this analysis. This analysis was completed for Adverse Event (AE) criteria related to pain and hypersensitivity (Pain, Pain in Extremity, Hypersensitivity, Hypersensitivity at implant site, Neuroma, and derivations of these descriptors) beginning after Operative Day (Operative Day+1). Revision surgeries for Pain-Related conditions documented as Ongoing were also included. Recovered/Resolved AEs were not included in the analysis unless the resolution was surgical revision. Unrelated AEs were also not included in this analysis. This is the Safety population which includes all subjects that received a nerve repair.
Time Frame: Operative Day+1, Month 1, Month 3, Month 6, Month 9, Month 12
Population: No interpolated data or modeling was used for this analysis. This is the Safety population which includes all subjects that received a nerve repair.
Measure: Count of Participants; unit: Participants
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 112 | 108
Participants | 2 | 9

9. Post Hoc Outcome: Analysis of Time to Recovery of Sensibility Measured By Static Two-Point Discrimination (Gaps 15-25 mm) (Data As-reported)
Description: A post-hoc analysis was performed to determine the difference between treatment groups in the time from index surgery to the recovery of sensibility in the target nerve repair. s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. Time to Recovery of sensibility is defined as the month of the subject's visit where they achieved s2PD of 2-15 mm and maintained s2PD through their last visit. Missing or incomplete assessments were not imputed. This analysis was completed on the Per Protocol population, defined as subjects with at least 6 months follow-up and no major protocol violations.
Time Frame: Assessed at Month 1, Month 3, Month 6, Month 9, Month 12
Population: No interpolated data or modeling was used for this analysis. This is the Per Protocol population which includes all subjects in baseline population who have completed a minimum of 6 months follow-up and have no major protocol violations. Results are a subset of the Per Protocol population by length of nerve gap for Month 1 to Month 12.
Measure: Mean (Full Range); unit: Months
Groups:
- Processed Nerve Allograft (PNA): Commercially available Processed Nerve Allograft for repair of nerve gap (nerve gaps 15-25 mm)
- Collagen Nerve Cuff: Commercially available collagen nerve cuff for repair of nerve gap (nerve gaps 15-25 mm)
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 35 | 33
Months | 3.0 [1 to 9] | 5.6 [1 to 12]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)

10. Post Hoc Outcome: Analysis of Time to Recovery of Sensibility Measured By Static Two-Point Discrimination by Nerve Gap Length (Gap Length 11-25mm) (Data As-reported)
Description: A post-hoc analysis was performed to determine the difference between treatment groups in the time from index surgery to the recovery of sensibility in the target nerve repair by gap length interval. Data were grouped by gap length, starting with 15-25 and incrementally including additional gap lengths (i.e. 14, 13, 12, 11, and 10) when statistical significance was observed between groups. s2PD is measured by blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. Time to Recovery of sensibility is defined as the month of the subject's visit where they achieved subject's achievement of s2PD of 2-15 mm and maintained s2PD through their last visit. This analysis was completed on the Per Protocol population, defined as subjects with at least 6 months follow-up and no major protocol violations.
Time Frame: Assessed at Month 3, Month 6, Month 9, and Month 12
Population: The failure to respond to stimulus was not recorded, thus only subjects with recovered sensibility are included in this data set. No interpolated data or modeling was used for this analysis. This is the Per Protocol population which includes all subjects in baseline population who have completed a minimum of 6 months follow-up and have no major protocol violations.
Measure: Mean (Full Range); unit: Months
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 57 | 53
Months | 4.4 [3 to 12] | 5.4 [3 to 12]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; p = 0.037, Wilcoxon (Mann-Whitney); This analysis was completed utilizing a one-sided Wilcoxon Rank Sum test

11. Post Hoc Outcome: Analysis of Recovered Sensibility Measured By Static Two-Point Discrimination by Nerve Gap Length (Gap Length 13-25mm) (Data As-reported)
Description: A post-hoc analysis was performed to determine the gap length (in mm) at which a statistically significant difference in the recovery of sensibility between treatment groups could be detected. Data were grouped by gap length, starting with 15-25 and incrementally including additional gap lengths (i.e. 14, 13 and 12) when statistical significance was observed between groups. s2PD is measured by a blinded assessor using a standardized discriminator tool that measures the innervation density and the subject's ability to discern between a single point and two distinct points between 2mm and 15mm. Patients with a result of 'absent' were not included in this analysis. This analysis was completed on the Per Protocol population, defined as subjects with at least 6 months follow-up and no major protocol violations. Data used for this analysis was from 6 months post-surgical follow-up to the date of each subject's latest completed s2PD assessment, whichever came last, assessed up to 12 months.
Time Frame: Up to Month 12
Population: No interpolated data or modeling was used for this analysis. As there is no pre-defined numerical value for absent response/failure in the data as-reported, patients with a result of 'absent' were not included in this analysis. This is the Per Protocol population which includes all subjects in baseline population who have completed a minimum of 6 months follow-up and have no major protocol violations.
Measure: Mean (Full Range); unit: mm of s2PD
Arm/Group | Processed Nerve Allograft (PNA) | Collagen Nerve Cuff
Number analyzed (Participants) | 48 | 43
mm of s2PD | 6.2 [2 to 14] | 7.6 [4 to 14]
Statistical Analysis 1: Comparison: Processed Nerve Allograft (PNA) vs Collagen Nerve Cuff; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney); One-sided Wilcoxon Rank Sum test was utilized for this analysis

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Processed Nerve Allograft | Collagen Nerve Cuff
All-Cause Mortality (participants affected / at risk) | 1/112 | 1/108
Serious Adverse Events (participants affected / at risk) | 6/112 | 2/108
Other Adverse Events (participants affected / at risk) | 12/112 | 15/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Processed Nerve Allograft (N=112) | Collagen Nerve Cuff (N=108)
Sickle cell anaemia with crisis - Unrelated (Blood and lymphatic system disorders) | 1 | 0 — Determined to be Unrelated to treatment
Acute kidney injury - Unrelated (Renal and urinary disorders) | 1 | 0 — Determined to be Unrelated to treatment
Staphylococcal bacteraemia - Unrelated (Infections and infestations) | 1 | 0 — Determined to be Unrelated to treatment
Retroperitonial haemorrhage - Unrelated (Gastrointestinal disorders) | 1 | 0 — Determined to be Unrelated to treatment
Septic shock - Unrelated (Infections and infestations) | 1 | 0 — Determined to be Unrelated to treatment
Embolic stroke - Unrelated (Hepatobiliary disorders) | 1 | 0 — Determined to be Unrelated to treatment
Deep vein thrombosis - Unrelated (Vascular disorders) | 1 | 0 — Determined to be Unrelated to treatment
Respiratory failure - Unrelated (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Determined to be Unrelated to treatment
Leukocytosis - Unrelated (Blood and lymphatic system disorders) | 1 | 0 — Determined to be Unrelated to treatment
Malignant hypertension - Unrelated (Vascular disorders) | 1 | 0 — Determined to be Unrelated to treatment
COVID-19 - Unrelated (Infections and infestations) | 1 | 0 — Determined to be Unrelated to treatment
Localized infection - Unrelated (Infections and infestations) | 1 | 0 — Determined to be Unrelated to treatment
Overdose - Unrelated (Injury, poisoning and procedural complications) | 1 | 0 — Determined to be Unrelated to treatment
Completed suicide - Unrelated (Psychiatric disorders) | 0 | 1 — Determined to be Unrelated to treatment
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 — Anticipated risk of a surgical procedure
Tendon rupture - Unrelated (Injury, poisoning and procedural complications) | 0 | 1 — Determined to be Unrelated to treatment
Cholecystitis - Unrelated (Hepatobiliary disorders) | 1 | 0 — Determined to be Unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Processed Nerve Allograft (N=112) | Collagen Nerve Cuff (N=108)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6
Implant site hypersensitivity (General disorders) | 3 | 5
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0

LIMITATIONS AND CAVEATS:
It is important to refer to the population being analyzed and the analysis methodology, as certain analyses include a repeated measures mixed modeling approach to address missing or incomplete data, while other analyses were conducted with as reported data. This resulted in certain populations containing extrapolated data for missing or incomplete data points and others excluded those subjects from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of at least sixty days prior to submission for publication for sponsor to review and comment. The Sponsor may extend the embargo for an additional 60 days to allow for the filing of a patent application or taking such measures Sponsor deems appropriate to establish and preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT01809002/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT01809002/SAP_001.pdf